CLINICAL TRIAL: NCT03240042
Title: Initial Increase in Cuff Pressure After Neck Retraction for Anterior Spine Surgery: Comparison Between Orotracheal and Nasotracheal Intubation
Brief Title: Initial Increase in Cuff Pressure in Anterior Cervical Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator, Associate Professor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-07-013C
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pressure Injury; Dysphonia; Dysphagia
Keywords: anterior cervical spine surgery; endotracheal cuff pressure; endotracheal tracheal intubation; dysphonia
MeSH Terms: conditions — Pressure Ulcer; Dysphonia; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated into one of the two group: nasoendotracheal and oroendotracheal group
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasoendo group (Experimental): Participants received nasotracheal intubation under general anesthesia for the anterior cervical spine surgery.
  Interventions: Procedure: nasotracheal intubation
- Oroendo group (Other): Participants received orotracheal intubation under general anesthesia for the anterior cervical spine surgery.
  Interventions: Procedure: orotracheal intubation

INTERVENTIONS:
Procedure: nasotracheal intubation — The participants either receive intubation via nasal route.
  Arms: Nasoendo group
Procedure: orotracheal intubation — The participants either receive intubation via oral route.
  Arms: Oroendo group

SUMMARY:
When the retractor blades oped and is positioned to provide the surgical access in the anterior cervical spine surgery, it cause the trachea to deviate laterally and pose pressure on the tissue between the retractor and the trachea. This is convincible as revealed by the increase of cuff pressure of endotracheal tube. The study aims to investigate differences in the increase of cuff pressure after retractor is positioned between nasotracheal and orotracheal intubation.

DETAILED DESCRIPTION:
When the retractor blades oped and is positioned to provide the surgical access in the anterior cervical spine surgery, it cause the trachea to deviate laterally and pose pressure on the tissue between the retractor and the trachea. The most important structure is the recurrent laryngeal nerve. This is convincible as revealed by the increase of cuff pressure of endotracheal tube. The pressure created by the retractor may be related to postoperative dysphonia and dysphagia. In view of minimizing the pressure created by the retractors, some neurosurgeons advocate to deflate then to inflate the cuff of ETT tube after the retractor is on, while some advocate monitoring of cuff pressure and keep below 25 mmHg. Nasotracheal or orotracheal tube can both be applied to general anesthesia for the anterior cervical spine surgery. The option depends on the surgeons' preference. Though both approaches end at the trachea, the nasotracheal tube is fixed at the nostril, and orotracheal tube, at the mouth angle, on the opposite side of surgical approach. The investigators hypothetize this difference in location results in different degree of deviation and increase of cuff pressure. The study aims to investigate differences in the increase of cuff pressure after retractor is positioned between nasoendotracheal and oroendotracheal intubation.

Apfelbaum and colleagues indicated the asymmetric position of the oroETT within the larynx as being fixed distally by the cuff and proximally by taping at the mouth angle. The asymmetry of the tube shaft and cuff may contribute to unilateral vocal palsy. When the retractors are set up for ACCS, the deviation of cuff towards the retractors increases ETCP and creates a extrusion compression of tissues in between the cuff and the retractor blade. Nasotracheal intubation follows a more natural trajectory into the trachea. In theory, a nasoETT is more centrally located and less asymmetric in the thyroid cartilage and trachea; thus pressure from this tube may be relatively evenly distributed, and the pressure on the surrounding tissues is lower. Therefore, we hypothesised lower degree of tissue compression with a nasoETT, even during retractor splay. The effect may be reflected in intraoperative ETCP or post-ACCS dysphonia. This randomised controlled clinical trial assessed the differences in the tracheal intubation mode on the maximal ETCP during retractor splay (primary endpoint) and post-ACSS dysphonia (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

Aged 20-80 Scheduled cervical spine surgery, anterior approach

Exclusion Criteria:

* Severe spinal stenosis and requiring fiberoptic intubation
* Unstable spine and require orthosis
* Hisotory of difficult intubation
* History of cervical spine or neck surgery
* Coagulopathy
* Nasal pathology
* Lack of informed consent
* History of previous cervical spine or neck surgery
* Anterior cervical spine surgeries after trauma, tumour resection, or spinal infection
* Preoperative dysphonia or dysphagia, regardless of the aetiology

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
cuff pressure | from time of randomization until postoperative 30 days
  cuff pressure of endotracheal tube

SECONDARY OUTCOMES:
sore throat | from time of randomization until postoperative 30 days
  postoperative sore throat by numerical rating scale (NRS), ranging from 0-10cm, 0 denoting minimal sore throat, 10 denoting maximal sore throat. score of 0 represents better outcome than score of 10.
dysphonia | from time of randomization until postoperative 30 days
  postoperative dysphonia by dysphonia scoring system. subjecte grading of voice change with none, mild and obvious, in terms of hoarseness,pitch and loudness.
dysphagia | rom time of randomization until postoperative 30 days
  postoperative dysphonia by BAZAZ dysphagia scoring system. Severity of dsyphagia is classified as none, mild, moderate and severe. None indicates no swallowing difficulty for liquid and solid food. Mild indicated no difficulty for liquid, and rare diffilulty for solid food. Moderate indicates none or rare difficulty for liquid, occasional difficulty for solid. Severe indicates presence of difficulty for liquid and frequent difficulty for solid food.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Cheng Huang, M.D.,Ph.D., Principal Investigator — Department of Neurosurgery, Neurological Institute
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang WC, Tan EC, Huang SS, Chou CJ, Chang WK, Chu YC. Postoperative Sore Throat Helps Predict Swallowing Disturbance on Postoperative Day 30 of Anterior Cervical Spine Surgery: A Secondary Exploratory Analysis of a Randomized Clinical Trial of Tracheal Intubation Modes. Dysphagia. 2022 Feb;37(1):37-47. doi: 10.1007/s00455-021-10247-x. Epub 2021 Feb 23. PMID 33620562